CLINICAL TRIAL: NCT04562753
Title: Clinical Trial to Estimate the Efficacy, Safety and Cost-utility of the Trapezium-Metacarpal (TMC) Prosthesis Compared to Suspensionplasty.
Brief Title: Clinical Trial to Estimate the Efficacy of the Trapezium-Metacarpal (TMC) Prosthesis Compared to Suspensionplasty.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació d'investigació Sanitària de les Illes Balears (Other Government)
Collaborators: Hospital Son Espases (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4144/20
Record Dates: First submitted 2020-08-19; First posted 2020-09-24 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: First CarpoMetacarpal Osteoartrithis; Basal Thumb Osteoartrithis
Keywords: CMC Prosthesis; CMC Arthroplasty; Suspensionplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Maïa® TMC Prosthesis (Lépine Groupe) (Active Comparator): Patients undergoing thumb basal joint arthroplasty using Maïa® TMC prosthesis as treatment of osteoarthritis.
  Interventions: Procedure: Maïa® TMC Prosthesis (Lépine Groupe)
- APL Suspensionplasty (Active Comparator): Patients undergoing thumb basal joint arthroplasty using APL Suspensionplasty as treatment of osteoarthritis.
  Interventions: Procedure: APL Suspensionplasty

INTERVENTIONS:
Procedure: Maïa® TMC Prosthesis (Lépine Groupe) — Patients undergoing thumb basal joint arthroplasty using Maïa® TMC prosthesis as treatment of osteoarthritis.
  Arms: Maïa® TMC Prosthesis (Lépine Groupe)
Procedure: APL Suspensionplasty — Patients undergoing thumb basal joint arthroplasty using APL Suspensionplasty as treatment of osteoarthritis.
  Arms: APL Suspensionplasty

SUMMARY:
The main objective of the study is to evaluate the efficacy, safety and cost-utility of the Trapezium-Metacarpal (TMC) prosthesis against Suspensionplasty with Abductor Pollicis Longus (APL) for the treatment of patients with first carpometacarpal (CMC) joint osteoarthritis (OA). Patients will be allocated to one of these two groups:

1. Maïa® TMC prosthesis (Groupe Lépine TM).
2. APL Supensionplasty

We will collect patient data using the questionnaires administeredat baseline and after the treatment. The primary outcome will be pain measured by visual analogue scale (VAS) and secondary outcomes will include health-related quality of life measured by EuroQuol 5D questionnaire,

DETAILED DESCRIPTION:
First Carpometacarpal joint osteoarthritis (CMC-OA) is a common problem, being the second location of degenerative osteoarthritis in the hand. The pain, weakness, and swelling cause considerable interference in the activities of daily living, especially in activities that involve repetitive fist-clamp movements.

The conservative treatment available (pain killers, physiotherapy and splints) do not always manage to achieve complete remission of the symptoms or prevent its recurrence. There are several surgical techniques to treat osteoarthritis of the first CMC. The most common surgical treatments used are prosthetic joint replacement and trapeziectomy. The later can be done as an isolated procedure or associated with tendon interposition, ligament reconstruction or both. The preference for indication for one treatment or another is based on personal experience rather than on the available studies, which are highly heterogeneous.

In addition, the direct and indirect costs (those associated with productivity losses as a result of sick leave from the perspective of society) associated with the use of a CMC prosthesis remain unknown, with the shorter recovery time being one of the reasons for its implantation.

The main objective of the study is to determine whether the trapeziometacarpal prosthesis is more effective, safe and cost-effective than suspension suspensionplasty. The secondary objective is to evaluate the functional outcome and estimate the indirect costs and the incremental cost-effectiveness and cost-utility (efficiency) ratios of the trapeziometacarpal prosthesis with respect to suspensionplasty as a treatment for osteoarthritis of the basal thumb joint.

The primary outcome will be measured using the Visual Analogue Scale (VAS). Secondary outcomes will include Quick-DASH and health-related quality of life measured using the European Quality of Life-5 Dimensions Questionnaire (EQ-5D) and. In addition, we will collect direct and indirect costs.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 or older.
* Diagnosis of First CMC OA.
* Non-responses to conservative treatment.
* Eaton Stage 2-3
* Physical and cognitive aptitudes to understand and give written informed consent.

Exclusion Criteria:

* Comorbidity with other medical conditions which would affect the hand (Carpal Tunnel Syndrome, De Quervain Tenosynovitis, Trigger Finger)
* Rheumatoid Arthritis
* Previous surgery in the same hand.
* Rejection to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Pain, pre- to post-operatively, as measured by a standard visual analogue score (VAS) diagram to grade perceived pain | Baseline, 3 weeks after surgery, 6 weeks after surgery, 3 months after surgery, 6 months, 1 year after surgery, 2 years after surgery
  The standard VAS diagram is a scale from 0 to 10 where 0 indicates No Pain (smiling face), and 10 indicates Worst possible, unbearable, excruciating pain (crying face).

SECONDARY OUTCOMES:
Health-related quality of life questionnaire Euro-Quol 5D (EQ-5D) | Baseline, 3 weeks after surgery, 6 weeks after surgery, 3 months after surgery, 6 months, 1 year after surgery, 2 years after surgery
  is a standardized instrument for measuring generic health status. It has been widely used in population health surveys, clinical studies, economic evaluation and in routine outcome measurement in the delivery of operational healthcare.
3 Change in Patient-Reported Function as measured by the short form Disabilities of the Arm, Shoulder, and Hand (QuickDASH) questionnaire, within and between procedure cohorts | Baseline, 3 weeks after surgery, 6 weeks after surgery, 3 months after surgery, 6 months, 1 year after surgery, 2 years after surgery
  The short form QuickDASH questionnaire will be completed as a reflection of patient-reported specific upper extremity function. Absolute improvement in QuickDASH score will be compared within groups longitudinally and between groups at each time point. QuickDASH scores range from 0 (no disability) to 100 (most severe disability)
Change in pre-operative pinch and grip strength as measured by kilograms of pressure. | Baseline, 3 weeks after surgery, 6 weeks after surgery, 3 months after surgery, 6 months, 1 year after surgery, 2 years after surgery
  Power grip using a Jamar (Jackson, MO) dynamometer, followed by lateral (key) and pulp-to-pulp pinch, will be recorded (both in kilograms) with a pinch meter, taking the greater strength of three successive attempts at each position with a 15 second rest between each attempt. The dynamic position of the thumb metacarpophalangeal (MCP) joint will be recorded with a small goniometer during lateral pinch testing (in degrees).
Direct and Indirect Costs | Baseline, 3 weeks after surgery, 6 weeks after surgery, 3 months after surgery, 6 months, 1 year after surgery, 2 years after surgery
  To estimate the costs of both interventions from the provider perspective, direct medical costs will be calculated using activity-based cost analysis.
  To estimate them from the perspective of society, indirect costs will be added to the direct costs, which will be calculated using the following variables: age, sex, educational level, employment status, profession. It is considered a reasonable measure of labor productivity is the remuneration in the labor market (average earnings or salary).
  The utility measure to be used in the cost-utility analysis is the quality-adjusted life years (QALY) as the utility measure. The profits will be obtained through the EQ-5D-5L instrument in its Spanish version and through rates validated for Spain.

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Salva-Coll, MD, PhD, Study Chair — Hospital Son Espases
Locations (1):
- Hospital Son Espases, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lirola-Palmero S, Salva-Coll G, Yanez-Juan AM, Sanchez-Iriso E. Cost-effectiveness and cost-utility of the ball-and-socket trapeziometacarpal prosthesis compared to trapeziectomy and ligament reconstruction: study protocol for a randomized controlled clinical trial. Trials. 2024 Mar 27;25(1):220. doi: 10.1186/s13063-024-08057-1. PMID 38532422